CLINICAL TRIAL: NCT04514146
Title: A Pilot Study on the Effects of Water-only Fasting and Refeeding on Body Composition and Insulin Resistance
Brief Title: The Effects of Water-only Fasting and Refeeding on Body Composition
Status: Completed | Type: Observational
Sponsor: TrueNorth Health Foundation (Other)
Responsible Party: Principal Investigator, Toshia Myers, Director, TrueNorth Health Foundation
Other Study IDs: TNHF2020-2VAT
Record Dates: First submitted 2020-08-12; First posted 2020-08-14 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Visceral Obesity; Insulin Resistance
Keywords: water-only fasting; HOMA-IR; insulin resistance; visceral adipose tissue
MeSH Terms: conditions — Obesity, Abdominal; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — sera and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Water-only Fasting Group: Overweight and obese, non-diabetic participants undergoing elective water-only fasting treatment
  Interventions: Other: Water-only fasting

INTERVENTIONS:
Other: Water-only fasting — In-patient water-only fasting for at least 10 days followed by at least 5 days of refeeding

SUMMARY:
This observational pilot study will assess the effects of water-only fasting on body composition and insulin resistance

DETAILED DESCRIPTION:
This pilot study will explore the effects of water-only fasting followed by an exclusively whole-plant-food diet free of added salt, oil, and sugar on body composition with a particular focus on visceral adipose tissue (VAT). The study will also extend a previous study assessing the effects of fasting and refeeding on Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) values and markers of cardiovascular health and inflammation by following participants for an additional 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Any gender
* 40-70 years old
* Fasting plasma glucose <126mg/dL and/or hemoglobin A1c <7%
* BMI between 25 and 40 kg/m2
* Elect and qualify for a water-only fast of at least 10 consecutive days
* Provide informed consent
* Internet and computer access
* Able to return for 6-week follow-up visit

Exclusion Criteria:

* Active malignancy
* Active inflammatory disorder including classic autoimmune connective tissue (Lupus, Sjogrens, ANCA), multiple sclerosis, and inflammatory bowel disorders (Ulcerative colitis, Crohn's)
* Stroke or heart attack within the last 12 months
* Break water-only fast before 10 days with juice or food.
* Break water-only fast after 10 days with juice or food before end-of-fast blood draw occurs.
* Leave center before completing at least 5 days of refeeding
* Unable to lay still on the back for at least 10 min
* Abdominal metal implants

Ages: 40 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Overweight and obese, non-diabetic participants chosen from voluntary patients
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Mean changes in visceral adipose tissue from baseline | Baseline, up to 10 to 40 days after baseline, up to 5 to 20 days after end of fast, 6-weeks after end of refeed
  Visceral adipose tissue will be estimated using Holigic Horizon dual-energy X-ray absorptiometry (DXA) machine and reported in grams

SECONDARY OUTCOMES:
Mean changes in total fat and lean mass and bone mineral content (BMC) from baseline | Baseline, up to 10 to 40 days after baseline, up to 5 to 20 days after end of fast, 6-weeks after end of refeed
  Total fat and lean mass and BMC will be estimated using Holigic Horizon dual-energy X-ray absorptiometry (DXA) machine and reported in grams

OTHER OUTCOMES:
Mean changes in lipid profile from baseline | Baseline, up to 10 to 40 days after baseline, up to 5 to 20 days after end of fast, 6-weeks after end of refeed
  Lipid profile will be assessed using serum to measure cholesterol, triglycerides, high-density lipoprotein (HDL), and lowdensity lipoprotein (LDL) and reported in mg/dL
Mean changes in weight from baseline | Baseline, up to 10 to 40 days after baseline, up to 5 to 20 days after end of fast, 6-weeks after end of refeed
  Weight will be measured on a digital scale and reported in kilograms (kg)
Mean changes in insulin resistance from baseline | Baseline, up to 10 to 40 days after baseline, up to 5 to 20 days after end of fast, 6-weeks after end of refeed
  Insulin resistance will be assessed using serum glucose and insulin to calculate homeostatic model of insulin resistance (HOMA-IR) [fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5]
Mean changes in abdominal circumference from baseline | Baseline, up to 10 to 40 days after baseline, up to 5 to 20 days after end of fast, 6-weeks after end of refeed
  Abdominal circumference will be measured on bare skin at the minimal waistline with a tension-sensitive, non-elastic tape and reported in centimeters (cm)
Mean changes in high sensitivity C-reactive protein (hs-CRP) from baseline | Baseline, up to 10 to 40 days after baseline, up to 5 to 20 days after end of fast, 6-weeks after end of refeed
  hsCRP will assessed using serum and reported in mg/L
Mean changes in Gamma-Glutamyl-Transferase (GGT) from baseline | Baseline, up to 10 to 40 days after baseline, up to 5 to 20 days after end of fast, 6-weeks after end of refeed
  GGT will assessed using serum and reported in U/L

CONTACTS AND LOCATIONS:
Overall Officials: Toshia R Myers, PhD, Principal Investigator — Director
Locations (1):
- Toshia Myers, Santa Rosa, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ibrahim MM. Subcutaneous and visceral adipose tissue: structural and functional differences. Obes Rev. 2010 Jan;11(1):11-8. doi: 10.1111/j.1467-789X.2009.00623.x. Epub 2009 Jul 28. PMID 19656312
- [Background] Tchkonia T, Thomou T, Zhu Y, Karagiannides I, Pothoulakis C, Jensen MD, Kirkland JL. Mechanisms and metabolic implications of regional differences among fat depots. Cell Metab. 2013 May 7;17(5):644-656. doi: 10.1016/j.cmet.2013.03.008. Epub 2013 Apr 11. PMID 23583168
- [Background] Unamuno X, Gomez-Ambrosi J, Rodriguez A, Becerril S, Fruhbeck G, Catalan V. Adipokine dysregulation and adipose tissue inflammation in human obesity. Eur J Clin Invest. 2018 Sep;48(9):e12997. doi: 10.1111/eci.12997. Epub 2018 Aug 3. PMID 29995306
- [Background] Shuster A, Patlas M, Pinthus JH, Mourtzakis M. The clinical importance of visceral adiposity: a critical review of methods for visceral adipose tissue analysis. Br J Radiol. 2012 Jan;85(1009):1-10. doi: 10.1259/bjr/38447238. Epub 2011 Sep 21. PMID 21937614
- [Background] de Mutsert R, Gast K, Widya R, de Koning E, Jazet I, Lamb H, le Cessie S, de Roos A, Smit J, Rosendaal F, den Heijer M. Associations of Abdominal Subcutaneous and Visceral Fat with Insulin Resistance and Secretion Differ Between Men and Women: The Netherlands Epidemiology of Obesity Study. Metab Syndr Relat Disord. 2018 Feb;16(1):54-63. doi: 10.1089/met.2017.0128. Epub 2018 Jan 17. PMID 29338526
- [Background] Patel P, Abate N. Body fat distribution and insulin resistance. Nutrients. 2013 Jun 5;5(6):2019-27. doi: 10.3390/nu5062019. PMID 23739143
- [Background] Moon HU, Ha KH, Han SJ, Kim HJ, Kim DJ. The Association of Adiponectin and Visceral Fat with Insulin Resistance and beta-Cell Dysfunction. J Korean Med Sci. 2018 Dec 26;34(1):e7. doi: 10.3346/jkms.2019.34.e7. eCollection 2019 Jan 7. PMID 30618514
- [Background] Gutch M, Kumar S, Razi SM, Gupta KK, Gupta A. Assessment of insulin sensitivity/resistance. Indian J Endocrinol Metab. 2015 Jan-Feb;19(1):160-4. doi: 10.4103/2230-8210.146874. PMID 25593845
- [Background] Gast KB, Tjeerdema N, Stijnen T, Smit JW, Dekkers OM. Insulin resistance and risk of incident cardiovascular events in adults without diabetes: meta-analysis. PLoS One. 2012;7(12):e52036. doi: 10.1371/journal.pone.0052036. Epub 2012 Dec 28. PMID 23300589
- [Background] Ormazabal V, Nair S, Elfeky O, Aguayo C, Salomon C, Zuniga FA. Association between insulin resistance and the development of cardiovascular disease. Cardiovasc Diabetol. 2018 Aug 31;17(1):122. doi: 10.1186/s12933-018-0762-4. PMID 30170598
- [Background] King LK, March L, Anandacoomarasamy A. Obesity & osteoarthritis. Indian J Med Res. 2013;138(2):185-93. PMID 24056594
- [Background] Utzschneider KM, Van de Lagemaat A, Faulenbach MV, Goedecke JH, Carr DB, Boyko EJ, Fujimoto WY, Kahn SE. Insulin resistance is the best predictor of the metabolic syndrome in subjects with a first-degree relative with type 2 diabetes. Obesity (Silver Spring). 2010 Sep;18(9):1781-7. doi: 10.1038/oby.2010.77. Epub 2010 Apr 8. PMID 20379148
- [Background] Jee SH, Kim HJ, Lee J. Obesity, insulin resistance and cancer risk. Yonsei Med J. 2005 Aug 31;46(4):449-55. doi: 10.3349/ymj.2005.46.4.449. PMID 16127767
- [Background] Merlotti C, Ceriani V, Morabito A, Pontiroli AE. Subcutaneous fat loss is greater than visceral fat loss with diet and exercise, weight-loss promoting drugs and bariatric surgery: a critical review and meta-analysis. Int J Obes (Lond). 2017 May;41(5):672-682. doi: 10.1038/ijo.2017.31. Epub 2017 Feb 2. PMID 28148928
- [Background] Chaston TB, Dixon JB. Factors associated with percent change in visceral versus subcutaneous abdominal fat during weight loss: findings from a systematic review. Int J Obes (Lond). 2008 Apr;32(4):619-28. doi: 10.1038/sj.ijo.0803761. Epub 2008 Jan 8. PMID 18180786
- [Background] Gomez-Arbelaez D, Bellido D, Castro AI, Ordonez-Mayan L, Carreira J, Galban C, Martinez-Olmos MA, Crujeiras AB, Sajoux I, Casanueva FF. Body Composition Changes After Very-Low-Calorie Ketogenic Diet in Obesity Evaluated by 3 Standardized Methods. J Clin Endocrinol Metab. 2017 Feb 1;102(2):488-498. doi: 10.1210/jc.2016-2385. PMID 27754807
- [Background] Freedland ES. Role of a critical visceral adipose tissue threshold (CVATT) in metabolic syndrome: implications for controlling dietary carbohydrates: a review. Nutr Metab (Lond). 2004 Nov 5;1(1):12. doi: 10.1186/1743-7075-1-12. PMID 15530168
- [Background] Romano L, Marchetti M, Gualtieri P, Di Renzo L, Belcastro M, De Santis GL, Perrone MA, De Lorenzo A. Effects of a Personalized VLCKD on Body Composition and Resting Energy Expenditure in the Reversal of Diabetes to Prevent Complications. Nutrients. 2019 Jul 4;11(7):1526. doi: 10.3390/nu11071526. PMID 31277506
- [Background] Liu FX, Flatt SW, Nichols JF, Pakiz B, Barkai HS, Wing DR, Heath DD, Rock CL. Factors Associated with Visceral Fat Loss in Response to a Multifaceted Weight Loss Intervention. J Obes Weight Loss Ther. 2017;7(4):346. doi: 10.4172/2165-7904.1000346. Epub 2017 Aug 14. PMID 29629240
- [Background] Johnstone AM. Fasting - the ultimate diet? Obes Rev. 2007 May;8(3):211-22. doi: 10.1111/j.1467-789X.2006.00266.x. PMID 17444963
- [Background] Shepherd JA, Ng BK, Sommer MJ, Heymsfield SB. Body composition by DXA. Bone. 2017 Nov;104:101-105. doi: 10.1016/j.bone.2017.06.010. Epub 2017 Jun 16. PMID 28625918
- [Background] Finnell JS, Saul BC, Goldhamer AC, Myers TR. Is fasting safe? A chart review of adverse events during medically supervised, water-only fasting. BMC Complement Altern Med. 2018 Feb 20;18(1):67. doi: 10.1186/s12906-018-2136-6. PMID 29458369